CLINICAL TRIAL: NCT01024738
Title: Study to Determine the Anti-plaque Efficacy of Commerical Toothpastes and an Oral Rinse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2008-PLA-05-RR
Record Dates: First submitted 2008-09-26; First posted 2009-12-03 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-10

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride toothpaste (Placebo Comparator): negative control toothpaste
  Interventions: Drug: Fluoride
- Triclosan/Fluoride toothpaste (Active Comparator): positive control toothpaste (Total toothpaste)
  Interventions: Drug: Triclosan, fluoride
- Chlorhexidine Oral Rinse (Active Comparator): positive control oral rinse
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Fluoride — Brush half mouth twice daily for four days.
  Arms: Fluoride toothpaste
Drug: Triclosan, fluoride — Brush twice daily
  Other Names: Total toothpaste
  Arms: Triclosan/Fluoride toothpaste
Drug: Chlorhexidine Gluconate — Rinse mouth twice a day
  Arms: Chlorhexidine Oral Rinse

SUMMARY:
Calibration study to determine the anit-plaque efficacy of commerical toothpastes and an oral rinse

DETAILED DESCRIPTION:
Training of new examiners and validation of new clinical site to run 4 day short-term plaque studies. All products are commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 to 65 years inclusive
* Have a minimum of 15 natural uncrowned teeth (excluding 3rd molars) present
* Give written informed consent
* Be in good general health
* No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the dental/medical professional monitoring the study
* If of childbearing potential and on birth control (Diaphragm, Birth Control Pills, Birth Control Implants, IUD (Intrauterine device), condoms)

Exclusion Criteria:

* Medical condition which requires pre-medication (antibiotics) prior to dental
* Visits/procedures
* Allergy to chlorhexidine
* Advanced periodontal disease (gum disease)
* 5 or more decayed, untreated dental sites (cavities)
* Diseases of the soft or hard oral tissues (gums or palate)
* Orthodontic appliances that interfere with plaque rating
* Abnormal salivary function
* Use of drugs that can affect currently salivary flow or production
* Use of antibiotics one (1) month prior to or during this study
* Use of any over the counter medications other than analgesics (i.e. aspirin, ibuprofen, acetaminophen,naproxyn)
* Pregnant or breastfeeding.
* Participation in another research study in the month preceding this study
* Allergic to common toothpaste or mouth rinse ingredients.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy) or individuals who have a high risk of infection from other causes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark LeFelt, DDS, Principal Investigator
Locations (1):
- TKL Research, Inc., Paramus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Performed at the clinic
Groups:
- Fluoride Toothpaste First: Fluoride toothpaste first,chlorhexidine oral rinse second, triclosan/fluoride last
- Triclosan/Fluoride Toothpaste First: triclosan/fluoride toothpaste first, fluoride toothpaste second, chlorhexidine oral rinse last
- Chlorhexidine Oral Rinse: chlorhexidine oral rinse first,triclosan/fluoride second, fluoride last
Period: First Intervention:
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Started | 7 | 7 | 8
Completed | 7 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Washout After 1st Intervention
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Started | 7 | 7 | 8
Completed | 7 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Second Intervention:
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Started | 7 | 7 | 8
Completed | 7 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Washout After 2nd Intervention
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Started | 7 | 7 | 8
Completed | 7 | 7 | 8
Not Completed | 0 | 0 | 0
Period: Third Intervention:
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Started | 7 | 7 | 8
Completed | 7 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Toothpaste: triclosan/fluoride toothpaste (positive control)
- Chlorhexidine Oral Rinse: chlorhexidine oral rinse (positive control)
- Total: Total of all reporting groups
Arm/Group | Fluoride Toothpaste | Total Toothpaste | Chlorhexidine Oral Rinse | Total
Number analyzed (Participants) | 7 | 7 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 8 | 22
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.23) | 50.5 (6.5) | 56.6 (5.5) | 50.43 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 20
  Male | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: Plaque score is Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: 4 Days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride Toothpaste | Total Toothpaste | Chlorhexidine Oral Rinse
Number analyzed (Participants) | 22 | 22 | 22
Units on a scale | 3.31 (0.48) | 3.31 (0.38) | 2.91 (0.36)
Statistical Analysis 1: Comparison: Fluoride Toothpaste vs Total Toothpaste vs Chlorhexidine Oral Rinse; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 2 month test period
Description: subjects used the product twice a day for 4 days with oral exams at beginning and end of treatment periods.
Arm/Group | Fluoride Toothpaste First | Triclosan/Fluoride Toothpaste First | Chlorhexidine Oral Rinse
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoride Toothpaste First (N=22) | Triclosan/Fluoride Toothpaste First (N=22) | Chlorhexidine Oral Rinse (N=22)
Non related adverse event (Social circumstances) | 0 (0) | 0 (0) | 1 (1) — subject reported a fracture in a tooth while eating white bread. Subject had the tooth repair with a composite filling. Subject continued with study without interuption. Event determined to be not related to study toothpaste or rinse use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days